CLINICAL TRIAL: NCT01647568
Title: Safety of Continuing Anti-platelet Agents During Colonoscopic Polypectomy: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda A Feagins, Staff Gastroenterologist, Dallas VA Medical Center
Other Study IDs: DVAMC-09-084
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Post-polypectomy Bleeding; Anti-platelet Therapy; Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Patients who are not on any anti-platelet/anti-coagulant therapy and present to our lab for a elective colonoscopy.
- Thienopyridine Users: Patients on Clopidogrel or prasugrel when they present for an elective colonoscopy.

SUMMARY:
At our VA hospital, in general, it is the policy of our GI lab to not stop our patients anti-platelet therapy whenever they see us for a routine colonoscopy. We do this because we believe the risk of stopping these sort of medications outweigh the risks of a complication from a colonoscopy.

Therefore, we are enrolling patients who are either on clopidogrel or prasugrel or not on any anti-platelet/anti-coagulant therapy that come to our GI lab routine colonoscopies. We perform the procedure just like we normally would and then follow-up with the patient 7 and 30 days after their procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the GI lab for elective colonoscopy

Exclusion Criteria:

* Patients on Coumadin or other anti-coagulants
* Patients with Inflammatory Bowel Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the GI lab for elective colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Feagins LA, Iqbal R, Harford WV, Halai A, Cryer BL, Dunbar KB, Davila RE, Spechler SJ. Low rate of postpolypectomy bleeding among patients who continue thienopyridine therapy during colonoscopy. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1325-32. doi: 10.1016/j.cgh.2013.02.003. Epub 2013 Feb 9. PMID 23403011